CLINICAL TRIAL: NCT05331651
Title: Effect of Glycopyrronium in Combination With Tropisetron in Anti-postoperative Nausea and Vomiting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Collaborators: Chongqing General Hospital (Other); Chongqing Medical University (Other); The People's Hospital of DAZU ，Chongqing (Unknown); The People's Hospital of Chongqing Kaizhou District (Unknown); Fuling Hospital affiliated to Chongqing University (Unknown); Qianjiang Central Hospital of Chongqing (Unknown); Stomatological Hospital of Chongqing Medical University (Unknown); People's Hospital of Changshou Chongqing (Unknown); The Ninth People's Hospital of Chongqing (Unknown); The First People's Hospital Of Chongqing Liang Jiang New Area (Unknown); People's Hospital of Xiushan County (Unknown); Wushan County People's Hospital (Unknown); Three Gorges Hospital of Chongqing University (Other); First Affiliated Hospital of Chongqing Medical University (Other); Department of Anesthesiology, Daping Hospital, Institute of Surgery Research, the Army Medical University (Unknown); The People's Hospital of Nanchuan (Unknown); Chongqing Traditional Chinese Medicine Hospital (Other); People's Hospital of Shapingba District， Chongqing (Unknown); Chongqing Liangping District People's Hospital (Unknown); Chongqing Jiangbei Hospital of Traditional Chinese Medicine (Unknown); People's Hospital of Chongqing Hechuan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Glycopyrronium in anti-PONV
Record Dates: First submitted 2022-04-11; First posted 2022-04-15 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2022-12

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Glycopyrrolate; Tropisetron; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glycopyrronium in Combination With Tropisetron (Experimental)
  Interventions: Drug: Glycopyrronium in Combination With Tropisetron
- Normal Saline in Combination With Tropisetron (Placebo Comparator)
  Interventions: Drug: Normal Saline in Combination With Tropisetron

INTERVENTIONS:
Drug: Glycopyrronium in Combination With Tropisetron — Glycopyrronium (0.2mg) in Combination With Tropisetron (4mg) intravenously given at the ending of the surgery.
  Arms: Glycopyrronium in Combination With Tropisetron
Drug: Normal Saline in Combination With Tropisetron — Normal Saline in Combination With Tropisetron (4mg) intravenously given at the ending of the surgery.
  Arms: Normal Saline in Combination With Tropisetron

SUMMARY:
To compare the anti-nausea and vomiting effect between glycopyrronium in combination with tropisetron and normal saline in combination with tropisetron for patients receiving elective surgery under general anesthesia. Based on this study the investigators intend to explore the feasibility of using glycopyrronium as adjuvant drug to prevent postoperative nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Non-cardiac surgery
* American Society of Anesthesiologists classification I-III
* Receive general anesthesia
* Voluntarily receive postoperative intravenous controlled analgesia

Exclusion Criteria:

* Puerpera or lactation women
* Allergy or existing contraindication to glycopyrronium and tropisetron
* Participate in other clinical drug trials within three months
* Can not follow with the study procedure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
incidence of postoperative nausea and vomiting | from the ending of surgery to 24 hours after surgery
  postoperative nausea and vomiting is recorded according to follow-up visits after surgery

SECONDARY OUTCOMES:
intensity of postoperative nausea | from the ending of surgery to 24 hours after surgery
  intensity of postoperative nausea is assessed using Numeric Rating Scale (0-10, 0 represents no uncomfortable felling, 10 represents tolerableness)
incidence of postoperative vomiting | from the ending of surgery to 24 hours after surgery
  postoperative vomiting is recorded according to follow-up visits after surgery
incidence of intervention requirement for nausea and vomiting | from the ending of surgery to 24 hours after surgery
  this event is recorded according to follow-up visits after surgery

OTHER OUTCOMES:
Postoperative pain intensity | from the ending of surgery to 24 hours after surgery
  Pain intensity is assessed by numerical rating scale (0-10, 0 represents painless; 10 represents intolerable pain)
Postoperative analgesic requirements | from the ending of surgery to 24 hours after surgery
  Analgesic requirements is assessed by recording the volume of patient controlled analgesia pump
degree of satisfaction | from the ending of surgery to 24 hours after surgery
  degree of satisfaction is assessed by patient using numerical rating scale (0-10, 0 represents unsatisfactory; 10 represents complete satisfaction)
adverse reaction related to glycopyrronium and ondansetron | from the ending of surgery to 24 hours after surgery
  adverse reaction is recorded according to follow-up visits after surgery

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, MD, Principal Investigator — The Second Affiliated Hospital, Chongqing Medical University
Locations (1):
- Department of Anesthesiology, The Second Affiliated Hospital, Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data for this study is available from the sponsor on reasonable request through email.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within five years

REFERENCES:
- [Derived] Chen J, Piao G, Luan G, Yu Y, Zheng W, Li Y, Zhang C, Duan Y, Zhao M, Zhang Y, Xiang W, Cheng L, Ji C, Duan G, Huang H. Effects of Glycopyrronium Bromide as an Adjuvant Treatment in the Prevention of Nausea and Vomiting After Abdominal, Thyroid, and Breast Surgery: A Multicenter Randomized Controlled Trial. Drug Des Devel Ther. 2025 Aug 19;19:7123-7134. doi: 10.2147/DDDT.S515670. eCollection 2025. PMID 40859968